CLINICAL TRIAL: NCT04544436
Title: A Phase IIIb Multicenter, Randomized, Double-blind, Controlled Study to Evaluate the Efficacy, Safety and Pharmacokinetics of a Higher Dose of Ocrelizumab in Adults With Relapsing Multiple Sclerosis
Brief Title: A Study to Evaluate the Efficacy, Safety and Pharmacokinetics (PK) of a Higher Dose of Ocrelizumab in Adults With Relapsing Multiple Sclerosis (RMS)
Acronym: MUSETTE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BN42082; 2020-000893-69 (EudraCT Number); 2023-506467-34-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2020-09-04; First posted 2020-09-10 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Multiple Sclerosis
Keywords: Relapsing Remitting Multiple Sclerosis; Higher Dose of CD20 Antibody Ocrelizumab; Efficacy, Safety and Pharmacokinetics
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting | interventions — ocrelizumab; Histamine Antagonists; Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ocrelizumab Higher Dose (Experimental): Participants will be randomized to receive a minimum of 5 higher treatment doses based on their body weight at baseline: 1200 mg (participant's body weight <75 kilograms [kg]) or 1800 mg (participant's body weight ≥ 75 kg) of ocrelizumab administered by IV infusion Q24W in the DBT phase. During the optional OLE phase, participants will continue with their assigned dose of ocrelizumab (either 1200 or 1800 mg) for approximately 96 weeks (4 doses in total). Mandatory methylprednisolone (or equivalent) and antihistaminic drug (e.g., diphenhydramine or equivalent) will be administered approximately 30-60 minutes prior to the start of each ocrelizumab infusion.
  Interventions: Drug: Ocrelizumab; Drug: Antihistamine; Drug: Methylprednisolone
- Ocrelizumab Approved Dose (Active Comparator): Participants will be randomized to receive a minimum of 5 treatment doses of 600 mg ocrelizumab administered by IV infusion Q24W in the DBT phase. During the optional OLE phase, participants will be offered a higher dose of ocrelizumab (either 1200 or 1800 mg), based on their body weight at OLE baseline, for approximately 96 weeks (4 doses in total). Mandatory methylprednisolone (or equivalent) and antihistaminic drug (e.g., diphenhydramine or equivalent) will be administered approximately 30-60 minutes prior to the start of each ocrelizumab infusion.
  Interventions: Drug: Ocrelizumab; Drug: Antihistamine; Drug: Methylprednisolone

INTERVENTIONS:
Drug: Ocrelizumab — The actual higher dose of ocrelizumab will be assigned to participants based on their body weight at baseline: 1200 mg (body weight <75 kg) or 1800 mg (body weight ≥ 75 kg). The first dose of ocrelizumab will be administered as two 600 mg or 900 mg IV infusions given 14 days apart. For the subsequent doses, ocrelizumab will be administered as a single 1200 mg or 1800 mg IV infusion Q24W. During the optional OLE phase, participants will continue with their assigned dose of ocrelizumab (either 1200 or 1800 mg) for approximately 96 weeks (4 doses in total).
  Other Names: Ocrevus
  Arms: Ocrelizumab Higher Dose
Drug: Ocrelizumab — Ocrelizumab will be administered at a dose of 600 mg Q24W. The first dose of ocrelizumab will be administered as two 300 mg IV infusions given 14 days apart. For the subsequent doses, ocrelizumab will be administered as a single 600 mg IV infusion Q24W.
  Other Names: Ocrevus
  Arms: Ocrelizumab Approved Dose
Drug: Antihistamine — Premedication with oral or IV antihistaminic drug (i.e., diphenhydramine 50 mg or an equivalent dose of an alternative) will be administered prior to each ocrelizumab infusion.
  Other Names: Non-Investigational Medicinal Product
Drug: Methylprednisolone — Premedication with 100 mg of methylprednisolone (or equivalent) will be administered by IV infusion prior to each ocrelizumab infusion.
  Other Names: Non-Investigation Medicinal Product

SUMMARY:
This is a randomized, double-blind, controlled, parallel group, multicenter study to evaluate efficacy, safety and PK of a higher dose of ocrelizumab per intravenous (IV) infusion every 24 weeks (Q24W) in participants with RMS, in comparison to the approved 600 milligrams (mg) dose of ocrelizumab.

DETAILED DESCRIPTION:
Participants will be treated for a minimum of 120 weeks in the double-blind treatment (DBT) phase. Upon positive primary results after the DBT phase, an optional higher dose extension treatment, open-label extension (OLE) phase is planned for eligible participants. The OLE will be carried out for approximately 96 weeks. Participants will be followed for safety for 48 weeks thereafter. Participants whose B-cell levels still did not replete to their baseline level or the low level of normal (LLN), whichever is lower, will move into the B-cell monitoring (BCM) phase following the safety follow-up phase. The study will end when all participants who were not treated with an alternative B-cell depleting therapy have repleted their B-cells to the baseline value or the LLN.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RMS
* At least two documented clinical relapses within the last 2 years prior to screening, or one clinical relapse in the year prior to screening. No relapse 30 days prior to screening and at baseline
* Participants must be neurologically stable for at least 30 days prior to randomization and baseline
* EDSS score, at screening and baseline, from 0 to 5.5 inclusive
* Average T25FWT score over two trials at screening and over two trials at baseline respectively, up to 150 (inclusive) seconds
* Average 9HPT score over four trials at screening and over four trials at baseline respectively, up to 250 (inclusive) seconds
* Documented magnetic resonance imaging (MRI) of brain with abnormalities consistent with MS at screening
* Participants requiring symptomatic treatment for MS and/or physiotherapy must be treated at a stable dose. No initiation of symptomatic treatment for MS or physiotherapy within 4 weeks of randomization
* Females of childbearing potential, agreement to remain abstinent or use adequate contraceptive methods
* Female participants without reproductive potential may be enrolled e.g. if post-menopausal or if surgically sterile

Exclusion Criteria:

* History of primary progressive MS at screening
* Any known or suspected active infection at screening or baseline (except nailbed infections), or any major episode of infection requiring hospitalization or treatment with IV antimicrobials within 8 weeks or treatment with oral antimicrobials within 2 weeks, prior to and during screening
* History of confirmed or suspected progressive multifocal leukoencephalopathy
* History of cancer, including hematologic malignancy and solid tumors, within 10 years of screening
* Immunocompromised state
* Receipt of a live or live-attenuated vaccine within 6 weeks prior to randomization
* Inability to complete an MRI or contraindication to gadolinium administration
* Contraindications to mandatory pre-medications for infusion-related reaction (IRRs)
* Known presence of other neurologic disorders that could interfere with the diagnosis of MS or assessments of efficacy and/or safety during the study
* Any concomitant disease that may require chronic treatment with systemic corticosteroids or immunosuppressants during the course of the study
* Significant, uncontrolled disease that may preclude participant from participating in the study
* History of or currently active primary or secondary, non-drug-related, immunodeficiency
* Pregnant or breastfeeding or intending to become pregnant
* Lack of peripheral venous access
* History of alcohol or other drug abuse within 12 months prior to screening
* Treatment with any investigational agent within 24 weeks prior to screening or treatment with any experimental procedure for MS
* Previous use of anti- cluster of differentiation 20 (CD20s) (including ocrelizumab), unless the last infusion was more than 2 years before screening, B-cell count is normal, and the stop of the treatment was not motivated by safety reasons or lack of efficacy
* Previous treatment with fingolimod, siponimod, or ozanimod within 6 weeks of baseline
* Previous treatment with natalizumab within 4.5 months of baseline
* Previous treatment with interferons beta (1a or 1b), or glatiramer acetate within 2 weeks of baseline
* Any previous treatment with mitoxantrone, cladribine, atacicept, alemtuzumab, and daclizumab - Previous treatment with any other immunomodulatory or immunosuppressive medication not already listed above without appropriate washout as described in the applicable local label. If the washout requirements are not described in the applicable local label, then the wash out period must be five times the half-life of the medication
* Any previous treatment with bone marrow transplantation and hematopoietic stem cell transplantation
* Any previous history of transplantation or anti-rejection therapy
* Treatment with IV immunoglobulin (Ig) or plasmapheresis within 12 weeks prior to randomization
* Systemic corticosteroid therapy within 4 weeks prior to screening
* Positive screening tests for active, latent, or inadequately treated hepatitis B
* Sensitivity or intolerance to any ingredient (including excipients) of ocrelizumab
* Any additional exclusionary criterion as per ocrelizumab local label, if more stringent than the above

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 864 (Actual)
Dates: Start 2020-11-26 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Time to Onset of 12-week Composite Confirmed Disability Progression (cCDP12) | Baseline up to approximately 4.3 years
  Time to onset of cCDP is defined as the first occurrence of a predefined confirmed progression event measured by Expanded Disability Status Scale (EDSS), Timed 25-foot Walk Test (T25FWT) or 9-hole Peg Test (9-HPT).

SECONDARY OUTCOMES:
Time to Onset of 24-week cCDP (cCDP24) | Baseline up to approximately 4.3 years
  Time to onset of cCDP is defined as the first occurrence of a predefined confirmed progression event measured by EDSS, T25FWT or 9-HPT.
Time to Onset of 48-week cCDP (cCDP48) | Baseline up to approximately 4.3 years
  Time to onset of cCDP is defined as the first occurrence of a predefined confirmed progression event measured by EDSS, T25FWT or 9-HPT.
Time to Onset of cCDP12 Independent of Protocol-defined Relapses (PDR) | Baseline up to approximately 4.3 years
  Time to onset of cCDP is defined as the first occurrence of a predefined confirmed progression event measured by EDSS, T25FWT or 9-HPT independent of PDR.
Time to Onset of 12-week Confirmed Disability Progression (CDP12) | Baseline up to approximately 4.3 years
  CDP, defined as a sustained increase from baseline in EDSS score of ≥1.0 point in participants with a baseline EDSS score of ≤5.5 or a sustained increase of ≥0.5 points in participants with a baseline EDSS score of >5.5.
Time to ≥ 20% Increase in 12-week Confirmed by T25FWT | Baseline up to approximately 4.3 years
  The T25FWT is a performance measure used to assess walking speed based on a timed 25-foot walk. The participant is directed to start at one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly and safely as possible.
Annual Rate of Percent Change From Baseline in Total Brain Volume | Baseline up to approximately 4.3 years
Time to 12-week Confirmed 4-point Worsening in Symbol Digit Modality Test (SDMT) | Baseline up to approximately 4.3 years
  The SDMT is a performance measure that has demonstrated sensitivity in detecting not only the presence of cognitive impairment but also changes in cognitive functioning over time and in response to treatment. Using a reference key, the examinee has 90 seconds to pair specific numbers with given geometric figures. Responses will be collected orally. A four-point change from baseline is typically considered clinically meaningful.
Time to 12-week Confirmed 8-point Increase in 12-item Multiple Sclerosis Walking Scale (MSWS-12) | Baseline up to approximately 4.3 years
  Self-reported measure of the impact of multiple sclerosis (MS) on the individual's ability to walk
Change in Neurofilament Light (NfL) at Week 48 for Participants Assigned to the Higher Dose Ocrelizumab Group | Baseline (Week 0), Week 48
  Biomarker for neurodegeneration NfL
Change in NfL at Week 48 for Participants Assigned to the Approved Dose Ocrelizumab Group | Baseline (Week 0), Week 48
  Biomarker for neurodegeneration NfL
Percentage of Participants With Adverse Events (AEs) | Baseline up to approximately 7.5 years
Serum Concentration of Ocrelizumab at Specified Time Points | Week 0, 2, 12, 24, 36, 48, 60, 72, 84, 96, 120
B-cell Levels in Blood | Baseline up to approximately 4.3 years
  Levels of blood B-cells is based on a highly sensitive assay that can accurately measure below 5 B-cells per microliter in blood
Percentage of Participants Achieving 5 or Less B-cells per Microliter of Blood | Baseline up to approximately 4.3 years
  Levels of blood B-cells is based on a highly sensitive assay that can accurately measure below 5 B-cells per microliter in blood
Change From Baseline in the Anti-drug Antibody (ADA) Levels | Week 0, 24, 48, 72, 96, 120

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (121):
- United States (25):
  - North Central Neurology Associates, Cullman, Alabama
  - Alabama Neurology Associates, Homewood, Alabama
  - 21st Century Neurology, Phoenix, Arizona
  - Profound Research, LLC, Carlsbad, California
  - Stanford University Medical Center, Stanford, California
  - Advanced Neurology of Colorado, LLC, Fort Collins, Colorado
  - Neurology Associates, PA, Maitland, Florida
  - University of South Florida, Tampa, Florida
  - American Health Network Institute, LLC, Avon, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - The NeuroMedical Clinic of Central Louisiana, Alexandria, Louisiana
  - Maine Medical Center, Scarborough, Maine
  - Dragonfly Research, LLC, Wellesley, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Cleveland Clinic Lou Ruvo, Las Vegas, Nevada
  - Dent Neurological Institute, Amherst, New York
  - UC Health Neurology, Dayton, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Abington Neurological Associates, Willow Grove, Pennsylvania
  - Tri-State Mountain Neurology, Johnson City, Tennessee
  - Hope Neurology, Knoxville, Tennessee
  - Bhupesh Dihenia M.D. P.A., Lubbock, Texas
  - Lone Star Neurology of San Antonio, San Antonio, Texas
  - Evergreen MS Center, Kirkland, Washington
- Argentina (3):
  - Centro de Especialidades Neurológicas y Rehabilitación - CENyR, Buenos Aires
  - CEMIC, Buenos Aires
  - Centro de Investigaciones Médicas Tucuman, San Miguel de Tucumán
- Austin Hospital, Heidelberg, Victoria, Australia
- Belgium (2):
  - Hospital Erasme, Brussels
  - Revalidatie en MS Centrum, Overpelt
- Brazil (4):
  - Instituto de Neurologia de Curitiba, Curitiba, Paraná
  - IMV Pesquisa Neurológica, Porto Alegre, Rio Grande do Sul
  - Clinica Neurologica, Joinville, Santa Catarina
  - CPQuali Pesquisa Clinica Ltda, São Paulo, São Paulo
- Canada (2):
  - Recherche Sepmus Inc., Greenfield Park, Quebec
  - Hotel-Dieu de Levis, Lévis, Quebec
- Rigshospitalet Glostrup, Glostrup Municipality, Denmark
- France (4):
  - Groupe Hospitalier Pellegrin, Bordeaux
  - CHU Hopital Gabriel Montpied, Clermont-Ferrand
  - CH St Vincent de Paul, Lille
  - Hôpital Charles Nicolle, Rouen
- Germany (8):
  - Charite - Universitätsmedizin Berlin, Berlin
  - St. Josef-Hospital, Klinik für Neurologie, Bochum
  - Universitätsklinikum "Carl Gustav Carus", Zentrum für Klinische Neurowissenschaften, Dresden
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Universität Leipzig, Leipzig
  - Universitätsklinikum Tübingen, Zentrum für Neurologie, Tübingen
  - Universitätsklinikum Ulm, Ulm
  - Deutsche Klinik für Diagnostik, Wiesbaden
- 401 Military Hospital of Athens, Athens, Greece
- Hungary (3):
  - S-Medicon Egeszsegugyi Szolgaltato Kft., Budapest
  - UNO Medical Trials Kft., Budapest
  - Somogy Vármegyei Kaposi Mór Oktató Kórház, Kaposvár
- Italy (7):
  - Universita? G. D'Annunzio, Chieti, Abruzzo
  - AOU Seconda Università degli Studi, Napoli, Campania
  - Policlinico Tor Vergata Dip. Neuroscienze-Clinica Neurologica-UOSD Sclerosi Multipla, Rome, Lazio
  - NCL Institute Neuroscience, Rome, Lazio
  - Policlinico Umberto I, Rome, Lazio
  - Fond. Istituto Neurologico C.Besta, Milan, Lombardy
  - IRCCS Istituto Neurologico Neuromed, Pozzilli, Molise
- Peru (6):
  - Hospital IV Alberto Sabogal Sologuren, Bellavista
  - Clinica Internacional, Lima
  - Instituto Nacional de Ciencias Neurológicas - Hospital Mogrovejo, Lima
  - Hospital Maria Auxiliadora, Lima
  - Hospital Nacional Dos de Mayo, Lima
  - Clinica Sanchez Ferrer, Trujillo
- Poland (14):
  - Neurocentrum Bydgoszcz sp. z o.o, Bydgoszcz
  - COPERNICUS Podmiot Leczniczy Sp. z o. o. Szpital im. M. Kopernika, Gdansk
  - MA-LEK Clinical Sp. Z o.o., Katowice
  - SPZOZ Uniwersytecki Szp. Klin. nr1 im.N.Barlickiego UM, Lodz
  - Centrum Neurologii Krzysztof Selmaj, Lodz
  - Indywidualna Praktyka Lekarska Prof. Dr Hab. N. Med. Konrad Rejdak., Lublin
  - Neurologiczny Niepubliczny ZOZ Centrum Leczenia SM Osrodek Bada? Klinicznych, Plewiska
  - EMC Instytut Medyczny SA, Późna
  - Nmedis sp. z o.o., Rzeszów
  - Osrodek Badan Klinicznych Euromedis, Szczecin
  - Centrum Medyczne NeuroProtect, Warsaw
  - Klinika Neurologii I Wydzialu Lekarskiego WUM w Warszawie, Warsaw
  - Instytut Psychiatrii i Neurologii II Klinika Neurologiczna, Warsaw
  - Wojskowy Instytut Medyczny - Pa?Stwowy Instytut Badawczy, Warsaw
- Portugal (3):
  - Hospital de Braga, Braga
  - Centro Hospitalar de Lisboa Ocidental - Hospital Egas Moniz, Lisbon
  - Hospital de Santa Maria, Lisbon
- Russia (14):
  - FSBHI Siberian Clinical Center of the Federal Medical and Biological Agency, Krasnoyarsk, Krasnoyarsk Krai
  - Neiro Clinica LLC, Moscow, Moscow Oblast
  - Research Center of Neurology of RAMS, Moscow, Moscow Oblast
  - Federal center of brain research and neurotechnologies, Moskva, Moscow Oblast
  - City Clinical Hospital #24, Moskva, Moscow Oblast
  - National Center of Social Significant Disease, Saint Petersburg, Sankt-Peterburg
  - N.P. Bechtereva Institute of the Human Brain, Saint Petersburg, Sankt-Peterburg
  - City Hospital #40 of Kurortniy Administrative District, Saint Petersburg, Sankt-Peterburg
  - SHI Sverdlovsk Regional Clinical Hospital #1, Yekaterinburg, Sverdlovsk Oblast
  - Vertebronevrologiya LLC, Kazan', Tatarstan Republic
  - KSMU Interregional Clinical Diagnostic Centre, Kazan', Tatarstan Republic
  - Ulyanovsk Regional Clinical Hospital, Ulyanovsk, Ulyanovsk Oblast
  - Saratov State Medical University of RosZdrav, Saratov
  - Nebbiolo Center for Clinical Trials, Tomsk
- Spain (6):
  - Complejo Hospitalario Universitario A Coruña (CHUAC), A Coruña, LA Coruna
  - Hospital Quiron de Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Alvaro Cunqueiro, Vigo, Pontevedra
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Puerta del Mar, Cadiz
  - Hospital Regional Universitario de Malaga ? Hospital General, Málaga
- Switzerland (3):
  - Universitätsspital Basel Medizin Neurologie, Basel
  - Inselspital Bern Medizin Neurologie, Bern
  - Ospedale Regionale di Lugano - Civico, Lugano
- Kocaeli University Hospital, Kocaeli, Turkey (Türkiye)
- Ukraine (12):
  - 5th Cherkasy City Center of Primary Health Care, Cherkasy
  - Mun.Med.Proph.Inst.?Chernihiv Reg.Hosp.?, Chernihiv
  - Bukovinsky SMU RMI Chernivtsi RCH, Chernivtsi
  - SI USSRI of Medical and Social Problems of Disabilities of MOHU, Dnipro
  - Regional Clinical Hospital, Ivano-Frankivsk
  - Municipal Nonprofit Enterprise of Kharkiv Regional Council Regional Clinical Hospital, Kharkiv
  - St.In.Inst. of Neurol.Psych.and Narcol.of the AMSU, Kharkiv
  - Medical Center of Private Execution First Private Clinic, Kyiv
  - Medical Center Dopomoga Plus, Kyiv
  - Lvivska oblasna tsentralna likarnia, Lviv
  - LCC "Medical center "Unimed", Zaporizhzhia
  - Municipal Non-profit Enterprise Zaporizhzhya Regional Hospital Zaporizhzhya Regional Council, Zaporizhzhia
- Derriford Hospital, Plymouth, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).